CLINICAL TRIAL: NCT01350544
Title: Treatment Advocacy Intervention for HIV-Positive African Americans
Acronym: TA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Laura Bogart, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MD006058 (NIH); R01MD006058 (NIH)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: HIV
Keywords: HIV; Adherence; African American/Black; Disparities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-list control (No Intervention): Participants in the wait-list control group will not receive the intervention until after the 6-month follow-up assessment.
- treatment advocacy (Experimental): Treatment advocacy is a 24-week intervention with booster sessions, including a 4-week intensive intervention followed by a 20-week maintenance period. In the first 4 weeks, all participants receive 4 individual weekly 60-minute sessions and 1 group HIV education session. In the next 20 weeks, all participants receive booster sessions in weeks 12 and 20, and a counselor check-in phone call in week 8 regarding need for new referrals and adherence barriers. Participants who have not demonstrated good adherence (≥90%) during the prior 2 weeks receive ≤4 additional booster sessions at weeks 14, 16, 22, and 24. Clients receive additional linkage with AIDS Project Los Angeles' (APLA) social service programs, as necessary.
  Interventions: Behavioral: Treatment Advocacy

INTERVENTIONS:
Behavioral: Treatment Advocacy — Treatment advocacy is a 24-week intervention with booster sessions, including a 4-week intensive intervention followed by a 20-week maintenance period. In the first 4 weeks, all participants receive 4 individual weekly 60-minute sessions and 1 group HIV education session. In the next 20 weeks, all participants receive booster sessions in weeks 12 and 20, and a counselor check-in phone call in week 8 regarding need for new referrals and adherence barriers. Participants who have not demonstrated good adherence (≥90%) during the prior 2 weeks receive ≤4 additional booster sessions at weeks 14, 16, 22, and 24. Clients receive additional linkage with APLA's social service programs, as necessary.
  Other Names: treatment education
  Arms: treatment advocacy

SUMMARY:
The investigators hypothesize that participants in the treatment advocacy intervention will show significantly better HIV treatment adherence than will participants in the no-treatment (wait-list) control group.

DETAILED DESCRIPTION:
Compared to other races/ethnicities, African Americans with HIV have lower levels of engagement in care, are less likely to be on antiretroviral treatment (ART), and are more likely to delay care and ART initiation; those on ART are less likely to be adherent at high enough levels for the treatment to be effective. We propose to test an innovative, culturally relevant treatment advocacy (TA) intervention for African Americans with HIV that targets social, cultural, and structural issues contributing to poor HIV treatment behaviors. TA, which has been sustained in many community organizations throughout the HIV epidemic, has never been systematically evaluated. TA facilitates patient navigation through the medical system and provides tailored HIV treatment education and client-centered counseling to improve adherence and engagement in care. TA targets structural issues in healthcare and patients' lives by advocating to providers to improve patient-provider relationships, recommending changes in treatment and/or providers (if needed), and referring patients to mental health and social services. TA is particularly appropriate for African Americans with HIV, who may be mistrustful of providers: it can be conducted outside of the medical system in a safe, neutral community setting by individuals not associated with patients' healthcare. We developed a culturally relevant TA program that additionally discusses factors such as racism that undermine healthcare in Black communities, by acknowledging and directly addressing patients' medical mistrust and stigma as coping strategies that arise in response to oppression. The specific aims are to (1) conduct a randomized controlled trial to examine the effects of a culturally relevant TA program on adherence among African Americans with HIV; (2) identify culturally relevant mediators that explain the effects of treatment advocacy on antiretroviral treatment adherence among African Americans with HIV (e.g., improved behavioral adherence skills, coping with stress/discrimination, mental health, and patient satisfaction; lower levels of HIV misconceptions, internalized HIV stigma/homophobia, medical mistrust, and substance use); and (3) explore culturally relevant moderators of the effects of treatment advocacy on antiretroviral treatment adherence among African Americans with HIV (e.g., access to care, discrimination, incarceration, poverty, social support, spirituality, and trauma). A sample of 200 African Americans with HIV will be randomly assigned to a TA intervention or wait-list control group. Participants will complete surveys at screening, and at 3- and 6-months post-baseline, to assess pre-, intra-, and post-intervention effects on adherence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* self-identify as African American or Black
* client of APLA
* they are on ART and missed at least 1 dose in the past month
* they have a currently detectable or unknown HIV viral load (or have not had a viral load test within the last six months).

Exclusion Criteria:

* received treatment advocacy in last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Bogart, PhD, Principal Investigator — RAND
Locations (1):
- AIDS Project Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogart LM, Mutchler MG, McDavitt B, Klein DJ, Cunningham WE, Goggin KJ, Ghosh-Dastidar B, Rachal N, Nogg KA, Wagner GJ. A Randomized Controlled Trial of Rise, a Community-Based Culturally Congruent Adherence Intervention for Black Americans Living with HIV. Ann Behav Med. 2017 Dec;51(6):868-878. doi: 10.1007/s12160-017-9910-4. PMID 28432578
- [Derived] Wagner GJ, Bogart LM, Mutchler MG, McDavitt B, Mutepfa KD, Risley B. Increasing Antiretroviral Adherence for HIV-Positive African Americans (Project Rise): A Treatment Education Intervention Protocol. JMIR Res Protoc. 2016 Mar 29;5(1):e45. doi: 10.2196/resprot.5245. PMID 27025399

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Advocacy: Treatment advocacy is a 24-week intervention with booster sessions, including a 4-week intensive intervention followed by a 20-week maintenance period. In the first 4 weeks, participants receive 4 individual weekly 60-minute sessions and 1 group HIV education session. In the next 20 weeks, all participants receive booster sessions in weeks 12 and 20, and a counselor check-in phone call in week 8 regarding need for new referrals and adherence barriers. Participants who have not demonstrated good adherence (≥90%) during the prior 2 weeks receive ≤4 additional booster sessions at weeks 14, 16, 22, and 24. Clients receive additional linkage with APLA's social service programs, as necessary.
Period: Overall Study
Arm/Group | Wait-list Control | Treatment Advocacy
Started | 108 | 108
Completed | 85 | 86
Not Completed | 23 | 22
Not completed — Administrative Withdrawal | 0 | 1
Not completed — Death | 1 | 2
Not completed — Moved out of LA County | 2 | 2
Not completed — Medical Issues | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Incarceration | 1 | 0
Not completed — Lost to Follow-up | 18 | 15

BASELINE CHARACTERISTICS:
Population: One participant was administratively withdrawn from the intervention condition because it was found that she was ineligible (not on medications) after being randomized to the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-list Control | Treatment Advocacy | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (10.2) | 50.1 (10.0) | 48.6 (10.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 79 | 78 | 157
  Female | 24 | 27 | 51
  Transgender | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 101 | 101 | 202
  Unknown or Not Reported | 0 | 0 | 0
Income [Count of Participants; unit: Participants]
  None | 11 | 10 | 21
  >$0 - <$10K | 66 | 53 | 119
  $10K - $20K | 18 | 35 | 53
  >$20K - $30K | 10 | 8 | 18
  >$30K - $40K | 2 | 0.0 | 2
  Unknown | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  7th to 11th Grade | 17 | 23 | 40
  High School diploma or GED | 37 | 33 | 70
  Some college | 41 | 40 | 81
  College degree | 6 | 7 | 13
  Some graduate school | 3 | 4 | 7
  Graduate degree | 4 | 0.0 | 4
Housing Status [Count of Participants; unit: Participants]
  Rent/Own | 65 | 69 | 134
  Treatment facility | 9 | 2 | 11
  Subsidized / Sect. 8 | 8 | 8 | 16
  Friend / relative | 11 | 8 | 19
  Temporary or transitional | 9 | 13 | 22
  Homeless | 5 | 6 | 11
  Other | 1 | 1 | 2
Employment Status [Count of Participants; unit: Participants]
  Full time | 4 | 1 | 5
  Part time | 4 | 5 | 9
  Unemployed | 63 | 71 | 134
  Retired | 19 | 14 | 33
  Other | 18 | 17 | 35
Length of Time Diagnosed [Mean (Standard Deviation); unit: years] | 15.3 (8.8) | 15.5 (7.9) | 15.5 (8.3)
Viral Load [Count of Participants; unit: Participants] — Medical record value closest to baseline
  Participants
    Detectable | 41 | 30 | 71
    Undetectable (<200 copies) | 41 | 54 | 95
    Unknown | 26 | 23 | 49
CD4 Cell Count [Mean (Standard Deviation); unit: cells per microliter] — Population: These values are based on medical records data. We could only obtain medical records data for a subset of participants.
  cells per microliter
    number analyzed (Participants) | 83 | 84 | 167
    (all) | 534 (316) | 650 (343) | 593 (334)
Received HIV care in last 6 months [Count of Participants; unit: Participants]
  received HIV care | 103 | 102 | 205
  did not receive HIV care | 5 | 5 | 10
Sexual Orientation [Count of Participants; unit: Participants]
  Straight | 36 | 43 | 79
  Gay man | 50 | 42 | 92
  Gay woman | 1 | 3 | 4
  Bisexual | 16 | 16 | 32
  Not Sure | 1 | 2 | 3
  Other | 4 | 2 | 6
Ever Incarcerated [Count of Participants; unit: Participants]
  ever incarcerated | 58 | 59 | 117
  never incarcerated | 49 | 48 | 97
  Unknow | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: We used a repeated measures linear regression modeling continuous adherence with intervention, linear time, and their interaction, and demographic covariates. Continuous adherence is measured as average percentages of doses taken.
Time Frame: Baseline, 1.5 months, 3 months, 4.5 months, and 6 months
Measure: Mean (Standard Deviation); unit: Percentage of doses taken
Groups:
- Treatment Advocacy: Treatment Advocacy: Treatment advocacy is a 24-week intervention with booster sessions, including a 4-week intensive intervention followed by a 20-week maintenance period. In the first 4 weeks, all participants receive 4 individual weekly 60-minute sessions and 1 group HIV education session. In the next 20 weeks, all participants receive booster sessions in weeks 12 and 20, and a counselor check-in phone call in week 8 regarding need for new referrals and adherence barriers. Participants who have not demonstrated good adherence (≥90%) during the prior 2 weeks receive ≤4 additional booster sessions at weeks 14, 16, 22, and 24. Clients receive additional linkage with APLA's social service programs, as necessary. This description is subject to change after consideration by the community advisory board.
Arm/Group | Wait-list Control | Treatment Advocacy
Number analyzed (Participants) | 85 | 86
Percentage of doses taken
  Baseline | 77.96 (23.15) | 80.13 (21.74)
  1.5 month follow-up | 64.87 (33.88) | 76.13 (25.55)
  3 month follow-up | 63.44 (33.01) | 76.76 (24.60)
  4.5 month follow-up | 63.69 (32.08) | 79.17 (25.31)
  6 month follow-up | 56.50 (33.97) | 78.76 (22.46)
Statistical Analysis 1: Comparison: Wait-list Control vs Treatment Advocacy; We used generalized linear mixed models predicting adherence at baseline and 1.5-, 3-, 4.5-, and 6-months post-baseline, with intervention , time, interaction between intervention and time, medical and socio-demographic covariates, and baseline viral load. Sample size was determined with a power analysis assuming .80 power and an alpha level of .05 that would allow for detection of a small-to-medium effect size in adherence between arms; Test type: Superiority; p = .005, Mixed Models Analysis — a priori threshold for significance for p < .05; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.69 to 0.91]

ADVERSE EVENTS:
Arm/Group | Wait-list Control | Treatment Advocacy
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107
Other Adverse Events (participants affected / at risk) | 0/108 | 0/107

LIMITATIONS AND CAVEATS:
We did not assess long-term effects, as the 6-month follow-up assessment occurred immediately after the last booster session. In addition, we did not assess the effects of the intervention on viral suppression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No